CLINICAL TRIAL: NCT03680729
Title: Adapting and Pilot Testing a Behavioral Intervention to Incorporate Advances in HIV Prevention for Black Young MSM in Alabama
Brief Title: Pilot Testing a Behavioral Intervention to Incorporate Advances in HIV Prevention for Black Young MSM in Alabama
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Henna Budhwani, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 520558
Record Dates: First submitted 2018-09-17; First posted 2018-09-21 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: HIV/AIDS
Keywords: Prevention; HIV/AIDS; MSM; Alabama
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: aBSB is the adaptation of BSB. BSB a two part intervention to improve rates of community-based HIV testing and prevention education in black young MSM (YMSM). BSB was developed on Information Motivation Behavioral Skills (IMB) theory. The first part of BSB uses Motivational Interviewing in a culturally appropriate way to encourage participants to accept testing and return for test results. The second part is conducted after the participant has received his result, assuming it was not reactive and offers prevention education.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aBSB (Experimental): aBSB is the adaptation of BSB. BSB a two part intervention to improve rates of community-based HIV testing and prevention education in black young MSM (YMSM). BSB was developed on Information Motivation Behavioral Skills (IMB) theory. The first part of BSB uses Motivational Interviewing in a culturally appropriate way to encourage participants to accept testing and return for test results. The second part is conducted after the participant has received his result, assuming it was not reactive and offers prevention education.
  Interventions: Behavioral: Adapted Brothers Saving Brothers (aBSB)
- Street Outreach (Active Comparator): Standard street outreach was used as the control in the original BSB trial.
  Interventions: Behavioral: Standard Street Outreach

INTERVENTIONS:
Behavioral: Adapted Brothers Saving Brothers (aBSB) — This information is listed in the arm description.
  Arms: aBSB
Behavioral: Standard Street Outreach — This information is listed in the arm description.
  Arms: Street Outreach

SUMMARY:
The overall goal of this 5-year Mentored Research Scientist Development K01-Award is to support Henna Budhwani, PhD, MPH to become an independent implementation science investigator in the field of HIV prevention. The proposed project seeks to address the HIV crisis in Alabama, where rates of undiagnosed HIV in black young men who have sex with men (YMSM, 18-29 years) exceed 20%. This project will adapt and test a behavioral intervention to promote HIV rapid testing in the community, deliver culturally appropriate prevention education, offer sociostructural support, and refer eligible participants for pre-exposure prophylaxis (PrEP). Four training objectives are proposed that are in lockstep with three specific aims.

DETAILED DESCRIPTION:
This study was developed in the spirit of the K01 mechanism, thoughtfully linking training to research. The research study proposed in this K01-application includes the conduct of three specific aims that are aligned with four training objectives.

Objective 1 outlines an intensive training and mentoring plan on social theory including theories of intersectionality and emerging masculinities.

Objective 2 provides in-depth training on qualitative research methods including how to conduct focus groups, in-depth interviews, and qualitative data analysis. Aim 1, which will be conducted after Objective 2, is to elucidate experiences, beliefs, and predictors related to delivery and utilization of HIV testing and prevention services for black YMSM using qualitative research methods, namely in-depth interviews with HIV prevention and outreach staff, focus groups with black YMSM, and in-depth interviews with other members of key population sub-groups such as transgender women and black YMSM who are no longer on PrEP, to inform the adaptation of BSB. Aim 1 will include 6 focus groups with black YMSM to explore perceptions and experiences with testing, prevention services, and PrEP as these relate to the adaptation of the intervention (estimated N=36-48). Aim 1 will include in-depth interviews with transgender women, black YMSM who have not taken an HIV-test in the past 6-months, black YMSM who are on PrEP, and black YMSM who were on PrEP but are no longer on PrEP (estimated N=16-24). This first aim will also include in-depth interviews with HIV prevention and outreach staff to document inner and outer contexts of community-based testing and clinical settings (estimated N=10). Thematic coding and analysis methods will be used to elucidate ways in which the intervention will need to be modernized and revised to be culturally acceptable to the target population and to address locally relevant structural barriers.

Objective 3 provides robust training on how to scientifically and iteratively adapt HIV behavioral interventions using validated frameworks, such as intervention mapping. Aim 2 is to adapt the Brothers Saving Brothers (BSB) intervention to include two HIV prevention tools (rapid testing and PrEP), to address structural barriers, and to be acceptable to black YMSM in Alabama. In Aim 2, I will use intervention mapping, informed by Aim 1 data, to iteratively adapt BSB to include the aforementioned updates. Since BSB will require extensive revisions, I have selected an intervention development framework (rather than an adaptation model) to guide the scientific adaptation process. After each cycle, the adapted intervention will be shared with CBO outreach staff and black YMSM to solicit their feedback. I anticipate 2-4 iterations (adaptations).

Objective 4 offers methodical training and mentoring in the field of implementation science. Aim 3, which concludes the proposed research study and K01 project, is to conduct a hybrid type 1 effectiveness-implementation pilot study of the adapted intervention in which the investigators will a) assess acceptability and feasibility of the adapted BSB (aBSB); b) preliminarily estimate effects on HIV prevention outcomes; and c) collect data on real-world implementation. I will pilot-test aBSB with black YMSM in Alabama (N=60); half will be randomized to the control condition; half will receive aBSB. I will collect effectiveness data (including acceptability and feasibility) pre-intervention/control, immediately post-intervention/control, 3-months after initial contact, and 6-months after initial contact. Toward the end of the study-period, I will collect implementation data from staff interviewed in Aim 1 (N=10) and from study participants to assess how aBSB was experienced and internalized (N=12).

This rigorous project includes intensive training at UAB and from other prominent institutions that offer very specific training not found at UAB; comprehensive mentoring from senior HIV researchers with expertise in minority, youth, and MSM health; and a thoughtful research strategy that addresses a significant threat -- high rates of undiagnosed HIV and the lack of HIV prevention, including PrEP uptake -- in black YMSM in Alabama. The combination of the proposed mentoring and training with study findings will culminate in the candidates attainment of independence and the development of a full-scale R01 implementation science proposal to test the adapted intervention.

ELIGIBILITY:
Inclusion Criteria for Staff:

* Minimally 18 years and 0 months of age
* Interacts with youth routinely
* Conducts or supervises community outreach and community-based HIV testing
* English speaking
* Can read English text
* Able and willing to provide informed consent

Inclusion Criteria for youth participants:

* Youth aged 18 years, 0 months to 29 years, 11 months
* Identifies as Black (or African American)
* Identifies as biologically male
* Is sexually active with male partners (MSM)
* Hasn't taken an HIV test in 6-months
* Is not currently on PrEP
* English speaking
* Able and willing to provide informed consent

Exclusion Criteria:

• Does not meet inclusion criteria

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — For part of the study, tentatively, only males will be eligible.
Enrollment: 59 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2025-01-11 (Actual); Study Completion 2025-01-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham (UAB), Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
All data gathered during the proposed study will be available to all participating mentors, advisors, and institutions. This includes the University of Alabama at Birmingham (UAB), University of California, San Francisco (UCSF), Florida State University College of Medicine, Wayne State University, Birmingham AIDS Outreach, and Selma AIR. All participating mentors and advisors will be included as authors in the dissemination of study findings through peer-review journals, conferences, and other presentations. Since the study will not develop model organisms or genome data, no sharing plan has been included for these contingencies.

REFERENCES:
- [Result] Budhwani H, Kiszla BM, Outlaw AY, Oster RA, Mugavero MJ, Johnson MO, Hightow-Weidman LB, Naar S, Turan JM. Adapting a Motivational Interviewing Intervention to Improve HIV Prevention Among Young, Black, Sexual Minority Men in Alabama: Protocol for the Development of the Kings Digital Health Intervention. JMIR Res Protoc. 2022 Jul 13;11(7):e36655. doi: 10.2196/36655. PMID 35830245

RESULTS

PARTICIPANT FLOW:
Groups:
- Kings: aBSB (renamed to Kings) is the adaptation of BSB into a digital health intervention.
- Standard Counseling: Standard of care control
Period: Overall Study
Arm/Group | Kings | Standard Counseling
Started | 35 | 24
Completed | 30 | 17
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kings | Standard Counseling | Total
Number analyzed (Participants) | 35 | 24 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.8 (2.4) | 26.0 (2.4) | 25.3 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 35 | 24 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 24 | 59
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 24 | 59

OUTCOME MEASURES:

1. Primary Outcome: Acceptability as Assessed by Participant Self-rated Satisfaction With the Intervention
Description: Participants rate their satisfaction with the intervention by positive response to "I like this app," scale of 1-4. Scores across participants in each arm were averaged to produce a mean score. Higher scores indicate higher acceptability.
Time Frame: 36 months
Measure: Mean (Full Range); unit: mean score on this question
Arm/Group | Kings | Standard Counseling
Number analyzed (Participants) | 30 | 17
mean score on this question | 3.47 [1 to 4] | 3.19 [1 to 4]

2. Primary Outcome: Did the Study Participant Accept a Rapid HIV Test After the Delivery of the Kings or Standard Outreach Intervention?
Description: This information will be assessed by the return of an HIV test result.
Time Frame: 18 months
Population: Total number of participants in each arm, converted to percentage, who shared their HIV test results with the study team.
Measure: Count of Participants; unit: Participants
Arm/Group | Kings | Standard Counseling
Number analyzed (Participants) | 30 | 17
Participants | 24 | 13

3. Secondary Outcome: Did the Study Participant Secure a Prescription for PrEP?
Description: This information will be assessed through clinical records. If the clinic reports that a script was issued, the measure will be marked as yes. If the clinic reports that a script was not issued, this measure will be marked as no.
Time Frame: 6 months
Population: Total number of participants who verifiably secured a prescription for PrEP.
Measure: Number; unit: participants
Arm/Group | Kings | Standard Counseling
Number analyzed (Participants) | 30 | 17
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: There was no difference in definition.
Arm/Group | Kings | Standard Counseling
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/24
Other Adverse Events (participants affected / at risk) | 0/35 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT03680729/Prot_SAP_000.pdf